CLINICAL TRIAL: NCT04558255
Title: Plasma Biomarkers as a Non-invasive Approach for Early Diagnosis of Lung Cancer
Brief Title: A Preliminary Study on the Detection of Plasma Markers in Early Diagnosis for Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jun Wang, Director of the Thoracic Surgery Department, Peking University People's Hospital
Other Study IDs: PTHO1903
Record Dates: First submitted 2020-09-13; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: A machine-learning method which can robustly discriminate early-stage lung cancer patients from controls — In our study, we intend to integrate molecular features obtained through liquid biopsy and clinical data of lung cancer patients, and develop and prospectively validate a machine-learning method which can robustly discriminate early-stage lung cancer patients from controls.

SUMMARY:
Lung cancer is the most common cancer with the highest morbidity and mortality in the world. Stagement is closely related to the 5 years of survival rate of patients. The postoperative 5-year survival rate is above 90% for stage ⅠA lung cancer patients, while the 5-year survival rate of stage IV lung cancer patients is less than 5%. Therefore, early screening and diagnosis for lung cancer is a key method to reduce lung cancer mortality and prolong survival for patients.

At present, low-dose computed tomography (LDCT) is the most effective method for early detection of lung cancer. In addition to imaging examination, plasma tumor markers detection is also a common clinical detection method for tumor screening and postoperative monitoring.

Liquid biopsy is a non-invasive or minimally invasive method for testing blood or other liquid samples to analyze tumor-related markers including nucleic acids and proteins. Several studies have explored the detection of hot spot gene mutations, methylation and methylation changes of DNA, protein markers and autoantibodies in peripheral blood in lung cancer patients. Liquid biopsy has generally become the most popular field for early diagnosis of lung cancer.

Based above, it is necessary to combine multi-omics methods to improve the detection of early stage lung cancer. In our study, we intend to integrate molecular features obtained through liquid biopsy and clinical data of lung cancer patients, and develop and prospectively validate a machine-learning method which can robustly discriminate early-stage lung cancer patients from controls.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled patients are newly diagnosed patients
* In patients diagnosed as pulmonary nodules by imaging, benign and malignant conditions of the nodules are determined by postoperative pathology after surgical resection
* There is clear cancer stage information
* In addition to pulmonary nodules, there are no suspicious nodules of other organs
* No previous history of malignant tumor

Exclusion Criteria:

* Patients with a history of malignant tumor
* Patients with suspectednodules in other parts of the body at the time of diagnosis
* Patients who have previously received surgery, chemotherapy or radiotherapy for pulmonary lesions
* Patients with severe blood lipid in peripheral blood extracted which affects subsequent detection

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 500 cases will be enrolled including 100 cases of benign pulmonary nodules, 300 cases of stage I and II lung cancer, 100 cases of stage III lung cancer. All enrolled patients are newly diagnosed as pulmonary nodules by imaging, benign and malignant conditions of the nodules are determined by postoperative pathology after surgical resection. All clinacal data including cancer stage information are available.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Rates of malignant and benign pulmonary nodules measured by the postoperative pathology | 5 days after the surgery
  After the sugery of each patients with pulmonary nodules, we will get the clinicopathologic characteristics of the patients. Tumor stage and grade will be evaluated by us and rates of malignant and benign pulmonary nodules will be the primary outcome which we follow.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Wang, M.D., Study Director — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China